CLINICAL TRIAL: NCT07097168
Title: Evaluating Clinical Course in Coronary Artery Bypass Patients Using the WHOOP Fitness Band Heart Rate Variability Application.
Brief Title: Using WHOOP Fitness Band to Measure Heart Health Variability Before and After Surgery
Status: Withdrawn | Type: Observational
Why Stopped: Changes to study staffing and lack of coordinator support.
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00004109
Record Dates: First submitted 2025-05-28; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Bypass Graft; CABG; Heart Surgery; Heart Disease; Coronary Artery Disease; WHOOP; HRV; Heart Rate Variability
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to use the WHOOP device to measure heart rate variability (HRV) in patients with coronary artery disease (CAD) before and after they have CABG (coronary artery bypass graft) surgery. The main questions it aims to answer are:

* Can changes in HRV, measured by the WHOOP device, help predict how well patients with CAD will recover after CABG surgery?
* Can HRV changes during the hospital stay give doctors useful information about the patient's recovery?

Participants will:

* Wear the WHOOP device before and after their CABG surgery to measure HRV.
* Share their health information to help researchers see how changes in HRV are connected to recovery.

This study will help find out if the WHOOP device can be used as a medical tool to track recovery in patients with CAD after CABG surgery.

ELIGIBILITY:
Inclusion Criteria:

* 20 Years or older
* Coronary Artery Disease diagnosis
* Must be scheduled for isolated Coronary Artery Bypass Surgery

Exclusion Criteria: Participants will be excluded if they have the following;

* Acute heart failure
* Acute coronary syndrome (e.g. heart attack/myocardial infarction) in the last 3 months.
* Prior history of heart transplant
* Cardiac assist device (e.g., ventricular assist device, balloon pump)
* Current pacemaker
* Congenital heart disease
* Currently admitted and undergoing treatment for cardiac issues e.g., inotropes, etc,
* Atrial fibrillation
* Frequent premature ventricular complex
* Sinus node dysfunction
* Second and third-degree atrioventricular block
* Combined cardiac surgeries
* Unable to consent.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants for validation will come from the general population and will be allowed to come forward to the study team to express interest. Study team members will place flyers in public areas (e.g., waiting rooms) throughout the Tufts Medical Center campus. Flyers will contain contact information of the study team as well as a QR Code to a screening form for participants to fill out if they are interested in participating.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-06-11 (Estimated); Primary Completion 2026-01-11 (Estimated); Study Completion 2026-03-11 (Estimated)

PRIMARY OUTCOMES:
Change in Heart Rate Variability (HRV) Before and After CABG Surgery | - Pre-operative, Up to 1 hour before surgery (Measurement taken in the pre-op area) - Post-operative, Up to 1 day after surgery - 3 days prior to ICU discharge.
  The primary goal of this study is to assess how heart rate variability (HRV) changes in patients with coronary artery disease (CAD) before and after coronary artery bypass graft (CABG) surgery.

SECONDARY OUTCOMES:
Understanding correlation in HRV measurements taken immediately after surgery compared versus HRV measurements taken prior to hospital discharge. | Two HRV measurements taken for comparison; - Post-operative, Up to 1 day after surgery - 3 days prior to ICU discharge.
  The secondary aim of this study would be to associate this change in HRV with the patient's clinical course to establish HRV as a way to assess current patient status and to predict clinical course and outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick C Cobey, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share all collected IPD, including demographic information, clinical measurements, and outcomes data (e.g., heart rate variability, recovery progress, and post-surgery health status). This data will be available for researchers who request it, in accordance with a data-sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Bellenger CR, Miller DJ, Halson SL, Roach GD, Sargent C. Wrist-Based Photoplethysmography Assessment of Heart Rate and Heart Rate Variability: Validation of WHOOP. Sensors (Basel). 2021 May 20;21(10):3571. doi: 10.3390/s21103571. PMID 34065516
- [Background] Tiwari R, Kumar R, Malik S, Raj T, Kumar P. Analysis of Heart Rate Variability and Implication of Different Factors on Heart Rate Variability. Curr Cardiol Rev. 2021;17(5):e160721189770. doi: 10.2174/1573403X16999201231203854. PMID 33390146
- [Background] Lakusic N, Slivnjak V, Baborski F, Cerovec D. Heart Rate Variability after Off-Pump versus On-Pump Coronary Artery Bypass Graft Surgery. Cardiol Res Pract. 2009;2009:295376. doi: 10.4061/2009/295376. Epub 2009 Sep 1. PMID 19936115
- [Background] Van Thanh N, Hien NS, Son PN, Son PT. Pattern Changes in the Heart Rate Variability of Patients Undergoing Coronary Artery Bypass Grafting Surgery. Cardiol Res Pract. 2022 Apr 30;2022:1455025. doi: 10.1155/2022/1455025. eCollection 2022. PMID 35535246
- [Background] Evrengul H, Tanriverdi H, Kose S, Amasyali B, Kilic A, Celik T, Turhan H. The relationship between heart rate recovery and heart rate variability in coronary artery disease. Ann Noninvasive Electrocardiol. 2006 Apr;11(2):154-62. doi: 10.1111/j.1542-474X.2006.00097.x. PMID 16630090
- [Background] Miller DJ, Sargent C, Roach GD. A Validation of Six Wearable Devices for Estimating Sleep, Heart Rate and Heart Rate Variability in Healthy Adults. Sensors (Basel). 2022 Aug 22;22(16):6317. doi: 10.3390/s22166317. PMID 36016077
- [Background] Dimeling G, Bakaeen L, Khatri J, Bakaeen FG. CABG: When, why, and how? Cleve Clin J Med. 2021 May 3;88(5):295-303. doi: 10.3949/ccjm.88a.20115. PMID 33941604
- [Background] Cromwell J, Mitchell JB, Stason WB. Learning by doing in CABG surgery. Med Care. 1990 Jan;28(1):6-18. doi: 10.1097/00005650-199001000-00003. PMID 2404169
- [Background] Malakar AK, Choudhury D, Halder B, Paul P, Uddin A, Chakraborty S. A review on coronary artery disease, its risk factors, and therapeutics. J Cell Physiol. 2019 Aug;234(10):16812-16823. doi: 10.1002/jcp.28350. Epub 2019 Feb 20. PMID 30790284